CLINICAL TRIAL: NCT07220499
Title: Whole Food Plant-based Diet to Improve Outcomes in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Cancer Care (Other)
Responsible Party: Principal Investigator, Dorothy Tenney, Research, Pacific Cancer Care
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PCC-001
Record Dates: First submitted 2025-10-21; First posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
Keywords: whole food plant-based diet
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole Food Plant-based Diet (Experimental)
  Interventions: Other: Whole Food Plant-based Diet

INTERVENTIONS:
Other: Whole Food Plant-based Diet — 6-months of a predominately whole food plant-based diet

SUMMARY:
The purpose of this research is to determine if consuming a whole food plant-based diet for six months impacts outcomes in men with prostate cancer that have a rising prostate-specific antigen (PSA) level. The main questions it aims to answer are:

Does a whole-food plant-based impact PSA? Does a whole food plant-based diet impact risk factors associated with treatment for prostate cancer including LDL cholesterol, hemoglobin A1C, C-reactive protein?

Participants will be asked to attend twelve two-hour plant-based cooking and nutrition classes throughout a six-month period, consume a mostly whole food plant-based diet, provide blood samples, and complete three-day food journals to assess nutrient intake.

DETAILED DESCRIPTION:
Ten men with histologically or cytologically confirmed adenocarcinoma of the prostate will be recruited from local urologists and oncologists. Eligible participants will be asymptomatic with a rising PSA on at least two tests no more than 6 months apart. Participants will come from one of four categories: 1) early stage, not on therapy; 2) non-metastatic prostate cancer on therapy; 3) metastatic, not on therapy; 4) metastatic, on antiandrogen (i.e. leuprolide) therapy that is no longer effective.

Participants will attend 12 two-hour group educational sessions at Pacific Cancer Care over the course of 24 weeks to encourage increased consumption of whole plant foods including fruits, vegetables, legumes, nuts, seeds, and decreased consumption of processed and animal foods including refined carbohydrates, meat, seafood, eggs, and dairy. Strict elimination of animal foods will not be required allowing dietary flexibility.

Educational sessions will consist of a 1-hour presentation on various nutrition topics with an emphasis on the benefits of whole plant foods, a 30-minute cooking demonstration of a whole food plant-based meal and taste test, and a 30-minute discussion. Participants will be encouraged to bring one support person, preferably someone they share meals with such as a spouse, to the sessions. A booklet summarizing the information presented in the educational sessions, including whole food plant-based recipes, will be provided to participants and their support person. Participants will be provided with a "take-home" ingredient that was used to prepare the meal in class and organic produce boxes from weeks 1 through 9 and $20 gift cards for weeks 10 through 24.

The primary outcome will be change in PSA, which will be measured at baseline, 12 weeks, and 24 weeks. Secondary outcome measures will be assessed at baseline and 24 weeks including changes in nutrient intake as assessed by 3-day food journals, LDL cholesterol, hemoglobin A1C, and high sensitivity C-reactive protein. Insulin-like growth factor-1 and insulin-like growth factor binding protein-3 will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Males 45-99 years of age
* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Increasing PSA on at least 2 sequential tests not more than 6 months apart.
* Eastern Cooperative Oncology Group Performance Status Scale of 0 to 2
* Adequate organ and marrow function, based upon meeting all of the following laboratory criteria:

  * White blood cell count ≥ 2500/mm3 (≥ 2.5 GI/L)
  * Platelets ≥ 50,000/mm3 (≥ 100 GI/L) without transfusion
  * Hemoglobin ≥ 9 g/dL (≥ 90 g/L)
  * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin ≤ 2x upper limit of normal (or for subjects with Gilbert's syndrome direct bilirubin WNL) Serum albumin ≥ 2.8 g/dl
* Willingness and ability to comply with all study-related procedures
* Capable of understanding and complying with the protocol requirements and must have signed the informed consent document

Exclusion Criteria:

* Nut or legume allergy
* Currently consuming a vegetarian or vegan diet
* Concurrent participation in other nutrition or weight loss programs
* Expected changes in exercise patterns during the study period
* Active prostatitis
* Insulin-dependent or requiring diabetes mellitus
* Expected changes in chronic medications, including statins or oral diabetes medication during the study period (including a change in medication dosage)
* Expected radiation, chemotherapy, bone resorptive agents or anti-androgen within 2 months of beginning the diet intervention
* Known history of electrolyte imbalance or micronutrient deficiency, e.g., magnesium, cobalamin
* Ongoing use of warfarin anticoagulants
* Diagnosed, active inflammatory bowel disease
* Alcohol and/or drug abuse
* Psychiatric illnesses or social situations that would limit compliance with study requirements including the inability or lack of equipment to perform basic cooking tasks

Ages: 45 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 11 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Prostate Specific Antigen | 6 months

SECONDARY OUTCOMES:
LDL-cholesterol | 6 months
  mg/dL
Hemoglobin A1C | 6 months
  % of total hemoglobin
high sensitivity C-reactive protein | 6 months
  mg/L

OTHER OUTCOMES:
Plasma insulin-like growth factor 1 | 6 months
  ng/mL
Plasma insulin like growth factor binding protein 3 | 6 months
  ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: John Hausdorff, MD, Principal Investigator — Pacific Cancer Care
Locations (1):
- Pacific Cancer Care, Monterey, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF